CLINICAL TRIAL: NCT04587661
Title: Designing an Implementation Strategy for Delivering Routine Mental Health Screening and Treatment for Adolescents and Adults With Sickle Cell Disease
Brief Title: Designing an Implementation Strategy for Delivering Routine Mental Health Screening and Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to obtain the intended sample size.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Charles Jonassaint, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20070307; R34MH125152-01 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Sickle Cell Disease; Depression; Anxiety
MeSH Terms: conditions — Anemia, Sickle Cell; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- off-the-shelf digital CBT (Active Comparator): standard implementation strategy that has no content or references to SCD, chronic pain, or the unique challenges facing minority groups
  Interventions: Behavioral: off-the-shelf digital CBT
- adapted digital CBT (Experimental): has content or references to SCD, chronic pain, and the unique challenges facing minority groups
  Interventions: Behavioral: adapted digital CBT

INTERVENTIONS:
Behavioral: off-the-shelf digital CBT — Cognitive behavioral therapy for depression and anxiety
  Arms: off-the-shelf digital CBT
Behavioral: adapted digital CBT — Cognitive behavioral therapy for depression and anxiety for individuals from a minority group with SCD
  Arms: adapted digital CBT

SUMMARY:
African Americans living with chronic health conditions are more likely to experience depression and other mental health disorders than their healthy counterparts, and are more likely to experience severe depression than whites, but less likely to be diagnosed or receive treatment. One especially vulnerable group is patients with sickle cell disease (SCD), a genetic blood disorder that primarily affects people of African descent, many of whom live in disadvantaged circumstances and are cared for in under-resourced settings. SCD causes severe acute and chronic pain, end-organ damage, and early mortality. Patients transitioning from adolescence to adulthood (ages16-30) are at high risk for mental health disorders and suicide.

Using mobile technology, the investigators can provide high-quality, evidence-based behavioral mental health treatment that reaches patients in different settings. Digital cognitive behavioral therapy (CBT) is effective for treating depression and anxiety and can be brought to scale at low cost. Despite the promise of digital CBT, there are barriers to its widespread use, particularly in low-resource settings serving minorities. Qualitative data show that cultural factors-lack of relatability, representation, and perceived stigma regarding mental health treatment-limit engagement with digital CBT programs. Population-and setting-specific adaptations to interventions can lead to their successful implementation and wider use. The investigators will work with a digital CBT program to decrease stigma and make it more relatable and relevant to young adults with SCD, by devising changes to advertising and promotion, and tailoring communication with an integrated health coach, Aim 1: Use implementation science (ImS) and human-centered design methods to define the barriers to delivering routine mental health screening and digital CBT to adolescents and young adults with SCD. Aim 2: Rapidly iterate, test, and evaluate adaptations to the implementation strategy for a coach-enhanced digital mental health service. Aim 3: Demonstrate that a population-specific implementation strategy improves engagement with a digital CBT-based mental health service.

The investigators will capitalize on our mobile technology tools, interdisciplinary expertise, and community-based partnerships to investigate the implementation of digital CBT into low-resource clinics and community-based organizations serving adolescents and adults with sickle cell disease.

DETAILED DESCRIPTION:
African Americans living with chronic medical conditions are at high risk for depression and other mental health disorders yet are less likely to be diagnosed or receive treatment than their white counterparts. Left untreated, depression can increase disease severity and risk for mortality. One especially vulnerable group is patients with sickle cell disease (SCD), a genetic blood disorder that primarily affects people of African descent and disproportionately impacts those living in disadvantaged circumstances. Sickle cell causes severe acute and chronic pain, end-organ damage, and early mortality. In SCD, the transition from adolescence to adulthood is a tumultuous period, characterized by social vulnerability, increased medical complications, and high health care utilization. Young adults in this age group, 16-30, are at high risk for mental health disorders and suicide.

Using mobile technology, the investigators can provide high-quality, evidence-based behavioral mental health treatment that reaches patients in under-resourced settings. Digital cognitive behavioral therapy (CBT), also known as computerized CBT, is effective for treating depression and anxiety, and can be easily brought to scale at low cost. Several meta-analyses have found digital CBT effective for treating depression and anxiety in white adults. The investigators' group has shown in a large-scale trial that it is effective for treating these symptoms among African American patients at 22 primary care clinics. In two adult sickle cell clinics, the investigators have shown that routine mental health screening and digital CBT delivered as part of usual care can improve depressive symptoms and daily pain among adults with SCD. The investigators' group has also used this method to treat pain in pediatric SCD patients.

Gap in evidence: Despite the promise of digital CBT, there are barriers to widespread use of this technology, particularly in low-resource settings serving minorities. Studies using digital CBT often suffer from high attrition and poor adherence. In real-world settings, uptake is poor even when the service is offered free of charge. These limitations affect patients living with SCD. The investigators will modify how a digital CBT program for mental health is delivered to these patient sat the patient, provider, and organizational levels, by adding references and content representing SCD, chronic pain, and stressors unique to African Americans. The investigators believe this approach will radically improve the implementation of mental health screening and treatment in low-resource settings such as clinics and community organizations serving adolescents and adults with SCD, and similar communities.

Strategy and goals: Population-and setting-specific adaptations to interventions can lead to their successful implementation and wider use, yet no studies show how much adaptation is needed to effectively implement digital CBT in different settings. Qualitative data from The investigators' group and others show that cultural factors-lack of relatability, representation, and perceived stigma regarding mental health treatment-limit engagement with digital CBT programs. The investigators' proposal will devise changes to advertising, promotion, and health coach communications, that will decrease stigma and make digital CBT more relatable and relevant to young adults with SCD. The investigators hypothesize that low-cost adaptations to a digital CBT program will have better engagement than digital CBT with standard implementation strategy.

Aim 1: Use implementation science (ImS) and human-centered design methods to define the barriers to delivering routine mental health screening and digital CBT to adolescents and young adults with SCD. By leveraging ImS theory, models, and frameworks, The investigators will systematically collect and analyze qualitative data to define and understand the problem, stakeholder needs, and cultural barriers to routine mental health screening and treatment in SCD clinics and the community. Specifically, the investigators will use the Behavior Change Wheel as a validated method for identifying the appropriate behavior change and implementation strategies.

Aim 2: Rapidly iterate, test, and evaluate adaptations to the implementation strategy for a coach-enhanced digital mental health service. Based on findings from Aim 1, the investigators will systematically develop, test, and evaluate changes to how the CBT program is advertised/promoted, and introduced to patients and providers. The investigators will tailor the messages and multimedia content that health coaches send to patients.

Aim 3: Demonstrate that a population-specific implementation strategy improves engagement with a digital CBT-based mental health service. The investigators will recruit 40 adolescents and young adults with SCD (ages 16-30) and comorbid depression and randomize them to either the off-the-shelf digital CBT program and standard implementation strategy that has no content or references to SCD, chronic pain, or the unique challenges facing minority groups, to adapted digital CBT with a SCD-specific implementation approach.

Addressing mental health in SCD is a major step to delivering quality care and improving outcomes for this, and other hard-to-reach, minority populations. This study will generate the necessary data and infrastructure to conduct a large scale, R01-funded, multi-site pragmatic trial to determine how digital CBT can be used as an effective, low-cost, and scalable mental health treatment for adolescents and young adults with SCD.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of SCD (any genotype)
* report significant depression or anxiety symptoms (i.e., Patient Health Questionnaire [PHQ-9] or Generalized Anxiety Disorder Scale [GAD-7] > 4)

Exclusion Criteria:

* Unable to read English or understand the consent process
* Cognitively impaired adults as determined by their treating physician
* Any condition that in the opinion of the investigator would not allow the patient to continue on the study

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Jonassaint, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Results from research conducted under this project will be shared in several ways. Manuscripts will be submitted for publication in high-quality peer-reviewed journals, following the NIH Public Access Policy guidelines. Findings will be presented at relevant national conferences, public lectures, scientific institutions, and meetings.
  The study datasets will be archived and made available to qualified individuals after a period of exclusive use by the research teams and after publication of the primary manuscripts, following NIH guidelines. The investigators will invite other investigators to submit ancillary studies using the data from the pilot trial and will work with those investigators to foster additional research studies and manuscripts.
Supporting Information: Study Protocol
Time Frame: The data will be available within 12 months of the completion of the trial. There will be no end date for its availability.
Access Criteria: Investigators with approved Institutional Review Board (IRB) protocol can access the data.

REFERENCES:
- [Derived] Nikolajski C, O'Brien J, Nardo E, Szigethy E, Jonassaint C. Tailoring a Digital Mental Health Program for Patients With Sickle Cell Disease: Qualitative Study. JMIR Ment Health. 2023 Apr 6;10:e44216. doi: 10.2196/44216. PMID 37023443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT
Started | 11 | 10
Completed | 11 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.73 (6.00) | 20.7 (6.43) | 21.76 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 21
PHQ score [Mean (Standard Deviation); unit: units on a scale] — This scale measures depressive symptoms with nine statements indicating how participants felt over the last 2 weeks. The scale asks for each statement "how many days have you been bothered by any of the following problems?" and provides a likert scale response ranging from 0-3 [0(not at all)-1(several days)-2( More than half the time)- 3 (All the time)].
  units on a scale | 11.18 (6.57) | 13.1 (5.86) | 12.1 (6.16)
Pain [Mean (Standard Deviation); unit: units on a scale] | 5.27 (3.17) | 6.7 (1.34) | 5.95 (2.52)
SCD Efficacy [Mean (Standard Deviation); unit: units on a scale] | 30.27 (6.07) | 28 (5.48) | 29.19 (5.77)
GAD score [Mean (Standard Deviation); unit: units] | 9.27 (4.71) | 9.6 (6.83) | 9.43 (5.67)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of App Use
Description: A measure of participant engagement.
  {Number of times the app has been open per week}
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: App opening per week
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT
Number analyzed (Participants) | 11 | 10
App opening per week | 5.64 (5.37) | 8.50 (8.98)

2. Primary Outcome: Number of Lessons Completed
Description: A measure of participant engagement.
  {Total number of lesson completed over the 4 week period}
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Lesson completed
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT
Number analyzed (Participants) | 11 | 10
Lesson completed | 1.27 (1.62) | 7.1 (13.94)

3. Primary Outcome: Number of Interactions (Text/Phone) With Health Coaches
Description: A measure of participant engagement.
  {Average number of texts messages sent to their health coach over the treatment period}
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Average text sent per week
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT
Number analyzed (Participants) | 11 | 10
Average text sent per week | 2.09 (2.98) | 6.1 (6.87)

4. Secondary Outcome: Change in Baseline Pain Scale at 4 Weeks
Description: The Pain scale asks participants to rank their average pain over the previous 7 days. The minimum score is 0. Maximum score is 10. The higher the score, the more severe the pain.
  (Value at Baseline -Value at 4 weeks = total change of average pain from baseline)
Time Frame: Baseline vs 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT
Number analyzed (Participants) | 10 | 7
score on a scale | 4.2 (1.93) | 3.86 (3.08)

5. Secondary Outcome: Change in Baseline Patient Health Questionnaire (PHQ-9) at 4 Weeks
Description: A 9-item measure of depressive symptoms. The minimum score is 0. The maximum score is 27. The higher the total score, the more severe the depressive symptoms.
  (Value at Baseline- Value at 4 weeks - = total change of depressive symptoms from baseline)
Time Frame: Baseline vs 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT
Number analyzed (Participants) | 11 | 8
units on a scale | 10.09 (4.89) | 6.57 (4.39)

6. Secondary Outcome: Change in Baseline Generalized Anxiety Disorder Scale (GAD-7) at 4 Weeks
Description: A 7-item measure of anxiety. The minimum score is 0. The maximum score is 21. The higher the total score, the more severe the symptoms of anxiety.
  ( Value at Baseline - Value at 4 weeks ) = total change of average anxiety symptoms from baseline)
Time Frame: Baseline vs 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT
Number analyzed (Participants) | 11 | 7
score on a scale | 8.91 (4.81) | 3.14 (4.49)

ADVERSE EVENTS:
Time Frame: Data was collected for the duration of the study (4 weeks).
Arm/Group | Off-the-shelf Digital CBT | Adapted Digital CBT
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
The sample size was lower than originally expected for this study so we were unable to test for covariates; Difficulties with recruitment required that the eligibility criteria was widened part way through recruitment to increase the available population pool;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT04587661/Prot_SAP_ICF_000.pdf